CLINICAL TRIAL: NCT04736862
Title: The Impact of Continuous Non-invasive Blood Pressure Monitoring on Post-induction and Intraoperative Hypotension in Patients Having Non-cardiac Surgery (DETECT Trial): A Randomized Trial
Brief Title: Impact of Continuous Non-invasive Blood Pressure Monitoring on Hypotension in Patients Having Non-cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PV7361
Record Dates: First submitted 2021-01-31; First posted 2021-02-03 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Blood Pressure; Perioperative Hypotension

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous monitoring group (Experimental)
  Interventions: Device: Continuous non-invasive blood pressure monitoring
- Intermittent monitoring group (Active Comparator)
  Interventions: Device: Intermittent non-invasive blood pressure monitoring

INTERVENTIONS:
Device: Continuous non-invasive blood pressure monitoring — In patients randomized to the continuous monitoring group, continuous non-invasive finger-cuff blood pressure monitoring will be displayed on the patient monitor. The treating anesthesiologist will be blinded to intermittent blood pressure monitoring using upper-arm cuff oscillometry.
  Arms: Continuous monitoring group
Device: Intermittent non-invasive blood pressure monitoring — In patients randomized to the intermittent monitoring group, intermittent blood pressure monitoring using upper-arm cuff oscillometry will be displayed on the patient monitor. The treating anesthesiologist is blinded to continuous non-invasive finger-cuff blood pressure monitoring.
  Arms: Intermittent monitoring group

SUMMARY:
This is a randomized trial (1) investigating whether continuous non-invasive finger-cuff blood pressure monitoring reduces the area under a mean arterial pressure (MAP) of 65 mmHg within the first 15 minutes of anesthetic induction compared to intermittent blood pressure monitoring using upper-arm cuff oscillometry in patients having non-cardiac surgery; and (2) investigating whether continuous non-invasive finger-cuff blood pressure monitoring reduces the time-weighted average for MAP <65 mmHg during the intraoperative period compared to intermittent blood pressure monitoring using upper-arm cuff oscillometry in patients having non-cardiac surgery.

DETAILED DESCRIPTION:
not provided

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 45 years of age scheduled for elective non-cardiac surgery with general anesthesia are eligible for study inclusion if blood pressure monitoring using intermittent upper-arm cuff oscillometry is planned.

Exclusion Criteria:

* Emergency surgery,
* pregnancy,
* American Society of Anesthesiologists (ASA) physical status classification V or VI, blood pressure differences between the right and left arm of more than 20 mmHg, intraoperative invasive blood pressure monitoring, heart rhythms other than sinus rhythm.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Area under a MAP of 65 mmHg within the first 15 minutes of anesthetic induction between the intervention and the control group. | 15 min
Time-weighted average for MAP <65 mmHg during the intraoperative period between the intervention and the control group. | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Karim Kouz, M.D., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Department of Anesthesiology, Center of Anesthesiology and Intensive Care Medicine, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kouz K, Weidemann F, Naebian A, Lohr A, Bergholz A, Thomsen KK, Krause L, Petzoldt M, Moll-Khosrawi P, Sessler DI, Flick M, Saugel B. Continuous Finger-cuff versus Intermittent Oscillometric Arterial Pressure Monitoring and Hypotension during Induction of Anesthesia and Noncardiac Surgery: The DETECT Randomized Trial. Anesthesiology. 2023 Sep 1;139(3):298-308. doi: 10.1097/ALN.0000000000004629. PMID 37265355